CLINICAL TRIAL: NCT07195019
Title: Treatments for Improving Mood in Women
Brief Title: Women's Wellbeing Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1871144-2; K23AT011917 (NIH)
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Distress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Yoga and Mindful Self-Compassion (I-YMSC) training (Experimental): 12 weeks of I-YMSC training
  Interventions: Behavioral: Integrative Yoga & Mindful Self-Compassion training
- Women's Wellbeing Education (WWE) (Active Comparator): 12 weeks of group WWE
  Interventions: Behavioral: Women's Wellbeing Education

INTERVENTIONS:
Behavioral: Integrative Yoga & Mindful Self-Compassion training — Group Integrative Yoga & Mindful Self-Compassion training for women with a history of interpersonal violence exposure and distress
  Arms: Integrative Yoga and Mindful Self-Compassion (I-YMSC) training
Behavioral: Women's Wellbeing Education — Group women's wellbeing education for women with a history of interpersonal violence exposure and distress
  Arms: Women's Wellbeing Education (WWE)

SUMMARY:
Phase 2 is a randomized controlled trial of integrative yoga and mindful self-compassion program vs. women's wellbeing education for women with a history of interpersonal violence exposure and heightened distress.

DETAILED DESCRIPTION:
In Phase 2, the investigators will conduct a pilot randomized controlled trial (RCT) of 12 weeks of integrative yoga and mindful self-compassion training (I-YMSC) vs. 12 weeks of women's wellbeing education (WWE).

Participants will be women with a history of interpersonal violence exposure and heightened distress.

Participants will be randomized to Phase 2 groups of 12 weeks of I-YMSC or WWE. Forty-eight women will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Ages 18-65
3. Report having experienced interpersonal violence (defined to include all forms throughout the lifespan, confirmed with the Trauma History Questionnaire (THQ])
4. Report being distressed, defined by a score of >5 on the Kessler-6 screener
5. Speak and understand English well enough to understand questionnaires when they are read aloud
6. Have access to a telephone through owning one, a relative/friend, or an agency
7. Have access to a device that will support use of the video platform we are using to conduct assessments and for home practice yoga video sessions

Exclusion Criteria:

1. Inability to be physically active, determined by a score >1 on the Physical Activity Readiness Questionnaire (PAR-Q) and physician non-consent of participation
2. Planned surgery in next 6 months, as this would interfere with study participation
3. Pregnancy, as yoga should be modified for pregnancy

   Women who meet criteria for the following:
4. Current mania as determined by the Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND)
5. Lifetime history of psychotic disorders (DIAMOND)
6. Current probable severe substance use disorder (DIAMOND)
7. Current diagnosis of anorexia nervosa or history in past year (DIAMOND)
8. Moderate or high risk for suicide on the adapted Columbia Suicide Severity Rating Scale screen version-recent (C-SSRS) and/or endorsement of suicidal plan/intent in the past 3 months
9. Non-stable course of psychiatric treatments (medication, psychotherapy) for the last 8 weeks
10. Plan to move from the area in the next 6 months, as this may preclude study participation given enrollment timeframes
11. Self-report of experiencing intimate partner violence currently or within past six months (assessed by the Revised Conflict Tactics Scale 2 [R-CTS2]), as this would require a different type of intervention
12. Current weekly yoga practice or current participation in mindfulness-based programming, as these are the study interventions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Post intervention (month 3)
  Feasibility assessed based on number of participants who remained in the intervention (retention).
Feasibility of Intervention Measure | Post intervention (month 3)
  The Feasibility of Intervention Measure (FIM) construct comprises four items with each item measured on a 1-5 scale. The total score range is from 4-20. Higher scores indicate greater feasibility.
Intervention Appropriateness Measure | Post intervention (month 3)
  The Intervention Appropriateness Measure (IAM) construct comprises four items with each item measured on a 1-5 scale. The total score range is from 4-20. Higher scores indicate greater feasibility.
Acceptability of Intervention Measure | Post intervention (month 3)
  The Acceptability of Intervention Measure (AIM) comprises four items with each item measured on a 1-5 scale. The total score range is from 4-20. Higher scores indicate greater feasibility.
The Client Satisfaction Questionnaire (CSQ-8) | Post intervention (month 3)
  Satisfaction with treatment assessed with The Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is an 8-item measure with each item measured on a 1-4 scale, and total score range from 8-32. Higher scores indicate greater client satisfaction.
Systematic Assessment of Treatment-emergent Events-general Inquiry (SAFTEE) | Post intervention (month 3)
  Participant safety/adverse events will be measured using the SAFTEE. Participants will also be asked weekly if they experienced any injuries as a result of yoga.

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS-21) | Baseline to post intervention (month 3)
  Distress at Month 3. The DASS-21 is a 21-item measure with each item measured on a 0-3 scale, and total score conversion ranging from 0-63. Higher global scores indicate greater psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided